CLINICAL TRIAL: NCT03075501
Title: Drug Contextual Conditioning With in Humans: Causes and Consequences
Brief Title: Interactions Between Drug Effects and Environments II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Emma Childs, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2015-0075; R21DA033488-01A1 (NIH)
Record Dates: First submitted 2016-05-18; First posted 2017-03-09 (Actual); Results first posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Substance-Related Disorders
Keywords: drug cues
MeSH Terms: conditions — Substance-Related Disorders | interventions — Central Nervous System Stimulants; Hypnotics and Sedatives

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paired (Active Comparator): Individuals receive drug (stimulant, or sedative) on two separate occasions and placebo on two separate occasions. Individuals receive drug in only one room.
  Interventions: Behavioral: Paired; Drug: Stimulant or sedative; Drug: Placebo
- Unpaired (Other): Individuals receive drug (stimulant, or sedative) on two separate occasions and placebo on two separate occasions. Individuals receive drug in both rooms.
  Interventions: Drug: Stimulant or sedative; Drug: Placebo

INTERVENTIONS:
Behavioral: Paired — Drug conditioning is assessed by pairing drug administration with a given context.
  Other Names: Conditioned place preference
  Arms: Paired
Drug: Stimulant or sedative — CS+ for paired, CS0 for unpaired
Drug: Placebo — CS- for paired, CS0 for unpaired

SUMMARY:
The purpose of the study is to determine how associations between drugs and the places where they are experienced influence drug seeking, mood and acute drug responses.

DETAILED DESCRIPTION:
Learned associations between drug effects and the people, places, and paraphernalia (cues) linked with drug experiences are a major barrier to the treatment of drug addiction. These links are remarkably persistent and can cause relapse to drug taking even after long periods of abstinence. They are also key features in some of the foremost theories of addiction, yet there is little clinical evidence of how these associations are formed and how they come to profoundly control behavior. The long-term goal of this research is to understand how drug cues become powerfully linked with drug experiences and their influence on mood and behavior. In the proposed project, the investigators will use a de novo conditioning paradigm to examine the influence of drug contexts on drug seeking, mood and acute drug responses. The hypothesis is that drug-paired contexts gain motivational salience, induce approach, and alter acute subjective responses to the drug.This knowledge will lead to novel treatment strategies to counteract the effects of drug cues on mood and behavior, and also to prevent relapse.

ELIGIBILITY:
Inclusion Criteria:

* past use of stimulants
* bmi 19-26
* hormonal birth control for women

Exclusion Criteria:

* current or recent (Past year) history of major axis I disorder

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emma Childs, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (N=133) were enrolled in the study between November 2015 and May 2018. All procedures were completed at the Human Addiction Pharmacology Laboratory at the University of Illinois at Chicago.
Pre-assignment Details: Participants underwent screening procedures to exclude participants who did not meet the study eligibility criteria.
Period: Overall Study
Arm/Group | Paired | Unpaired
Started | 89 | 44
Completed | 74 | 35
Not Completed | 15 | 9
Not completed — Scheduling difficulties | 15 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paired | Unpaired | Total
Number analyzed (Participants) | 74 | 35 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.7 (5.0) | 25.0 (4.6) | 24.8 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 14 | 38
  Male | 50 | 21 | 71
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian | 2 | 0 | 2
  Race: Asian | 7 | 5 | 12
  Race: Black or African American | 6 | 7 | 13
  Race: White | 47 | 20 | 67
  Race: More than 1 | 11 | 3 | 14
  Race: Unknown | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 74 | 35 | 109

OUTCOME MEASURES:

1. Primary Outcome: Change in Time Spent in Drug-paired Room
Description: The amount of time spent in the two testing rooms is assessed during a 10min exploration test conducted at the orientation session (pre-test) and again at the testing session (post-test). Between the pre- and post-tests, participants complete 4 drug administration sessions; 2 with 20mg MA, 2 with 0mg MA. The Paired Group always receives 20mg MA in the room they spent the least time in at pre-test, and 0mg MA in the other room. The Unpaired Group receives 20mg MA and 0mg MA once in each room. The research question is whether the Paired Group spends significantly more time in the room paired with 20mg MA in comparison to the Unpaired Group. Thus, the outcome measure is the difference in time spent in the room paired with drug administration (i.e. the room that they spent the least time in at pre-test) between pre- and post-tests (i.e., post-test time spent - pre-test time spent) which is compared between the groups. NOTE: Time spent is NOT obtained during drug administration sessions.
Time Frame: Measured through study completion (maximum 5 weeks).
Population: Video recordings of the exploration tests (used to calculate time spent) were unavailable (corrupted) for at least one test (pre- or post-) for 3 Paired participants and 2 Unpaired participants. Thus, the participant numbers for this analysis are reduced in comparison to the total number of participants who completed the study.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Paired: Participants complete 4 drug administration sessions; 2 each with 20mg MA or 0mg MA (placebo).
  Paired: Participants always receive MA in the room that they spent the least time in at the pre-test exploration test, and placebo in the other room.
  MA: CS+ for paired, CS0 for unpaired Placebo: CS- for paired, CS0 for unpaired
- Unpaired: Participants complete 4 drug administration sessions; 2 each with 20mg MA or 0mg MA (placebo).
  Unpaired: Participants receive MA and placebo once in each room i.e., drug administration is not paired with a given room.
  MA: CS+ for paired, CS0 for unpaired Placebo: CS- for paired, CS0 for unpaired
Arm/Group | Paired | Unpaired
Number analyzed (Participants) | 71 | 33
seconds | 24.5 (115.5) | 6.2 (122.4)

2. Secondary Outcome: Subjective Drug Effects
Description: Self-reported drug effects are measured using standardized questionnaires 30min before capsule administration (baseline) and at 30min intervals after capsule administration for 4h during each drug administration session. The peak change from baseline is calculated for each session and averaged across drug and placebo sessions. A net difference is calculated by subtracting the mean peak change from baseline during placebo sessions from the mean peak change from baseline during drug (20mg MA) sessions.
  Outcome measure: Subjective stimulation (i.e., feeling alert, aroused, energetic) is measured using the Amphetamine scale of the Addiction Research Center Inventory. Scores range from 0-11 with greater scores indicating greater drug effects.
Time Frame: Self-reported drug effects are measured 30min before drug administration and at 30min intervals after drug administration for 4h during each drug administration session.
Population: Data was analyzed only for participants who had complete data for the primary outcome (time spent).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Unpaired: Participants complete 4 drug administration sessions; 2 each with 20mg MA or 0mg MA (placebo).
  Unpaired: Participants receive MA once in each room and placebo once in each room.
  MA: CS+ for paired, CS0 for unpaired Placebo: CS- for paired, CS0 for unpaired
Arm/Group | Paired | Unpaired
Number analyzed (Participants) | 71 | 33
units on a scale | 3.4 (2.5) | 4.1 (2.5)

ADVERSE EVENTS:
Time Frame: Up to 5 weeks
Description: Participants reported adverse effects during and after sessions.
Groups:
- 20mg Methamphetamine; 0mg Methamphetamine (Placebo): Participants completed two drug administration sessions with 20mg methamphetamine.
  Self-reported side effects: At 30min intervals following drug administration (for 4h), they reported any side effects on a paper and pencil form. Drug side effects (Blurred vision, Dry mouth, Headache, Nausea, Heart racing, Shortness of breath, Dizziness/faintness, Restlessness, Chest discomfort, Shakiness or trembling (legs, arms, hands, feet), Pain or numbness in fingers or toes, Anxiety/tension) were each associated with a 100mm visual analogue scale anchored at the left hand side with "None" and at the right hand side with "Extreme". Participants placed a vertical line bisecting the scale that corresponded with how they were feeling at that time. Scores ranged from 0-100, with higher scores indicating more severe side effects.
  Cardiovascular Measures: Heart rate (bpm) and blood pressure mmHg) were monitored using a monitor 30min before drug administration (baseline) and at 30min intervals (for 4h) following drug administration.
  Serious adverse events were defined as any side effects reported in the "severe-extreme" range (i.e., >60) or any occasion when the study physician was consulted about high cardiovascular measures.
  Serious adverse events are reported for all participants who completed the study (N=109).
Arm/Group | 20mg Methamphetamine | 0mg Methamphetamine (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/109
Serious Adverse Events (participants affected / at risk) | 11/109 | 2/109
Other Adverse Events (participants affected / at risk) | 0/109 | 0/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 20mg Methamphetamine (N=109) | 0mg Methamphetamine (Placebo) (N=109)
High heart rate and blood pressure (Cardiac disorders) | 1 | 0 — The physician was consulted on one occasion regarding high heart rate and blood pressure values in a participant after receiving 20mg MA. The participant reported no additional adverse effects and after resting, heart rate and blood pressure reduced.
Dry mouth (Nervous system disorders) | 6 | 1
Shakiness/Trembling (Nervous system disorders) | 2 | 0
Heart racing (Cardiac disorders) | 2 | 0
Dizziness/faintness (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT03075501/Prot_SAP_ICF_000.pdf